CLINICAL TRIAL: NCT02565186
Title: An Open-label, LonG-term, Safety Study of LAsmiDItan (100 mg and 200 mg) in the Acute Treatment Of MigRaine (GLADIATOR)
Brief Title: An Open-label, Long-term, Safety Study of Lasmiditan for the Acute Treatment of Migraine
Acronym: GLADIATOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: CoLucid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16890; H8H-CD-LAHL (Other: Eli Lilly and Company); 2015-005674-37 (EudraCT Number); COL MIG-305 (Other: Colucid)
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2019-11

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — lasmiditan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lasmiditan 100mg (Experimental): Participants received oral dose of 100 milligrams (mg) Lasmiditan with in four hours of onset of migraine attack. If the migraine did not respond within 2 hours after first dose or if responded and recurred then a second dose was permitted within 24 hours after first dose.
  Interventions: Drug: Lasmiditan
- Lasmiditan 200mg (Experimental): Participants received oral dose of 200mg Lasmiditan with in four hours of onset of migraine attack. If the migraine did not respond with in 2 hours after first dose or if responded and recurred then a second dose was permitted within 24 hours after first dose.
  Interventions: Drug: Lasmiditan

INTERVENTIONS:
Drug: Lasmiditan — oral tablet
  Other Names: LY573144

SUMMARY:
This is a prospective, randomized, open-label study in subjects with migraine who have completed the Phase 3 studies, COL MIG 301/LAHJ (NCT02439320) or COL MIG-302/LAHK (NCT02605174) or for a subset of lasmiditan-naïve subjects with migraine. The study is designed to evaluate the safety and tolerability of long-term intermittent use of lasmiditan 100 mg and of lasmiditan 200 mg, as the first dose and as a second dose, for the acute treatment of migraine. Long term efficacy will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent and authorize Health Insurance Portability and Accountability Act (HIPAA).
* Completed COL MIG-301 or COL MIG-302 within the last 12 weeks. Subjects that completed COL MIG-301 prior to COL MIG-305 being available will be allowed to enroll as long as enrollment occurs within 4 weeks of COL MIG-305 activation at their site. (NOTE: Additional subjects may qualify if they completed COL MIG-301 or COL MIG-302 >12 weeks prior or if they have not participated in either prior study, but meet eligibility criteria outlined for COL MIG-302.)
* Females of child-bearing potential must be using or willing to use a highly effective form of contraception (e.g. combined oral contraceptive, intrauterine device (IUD), abstinence or vasectomized partner).
* Able and willing to complete an electronic diary to record details of all migraine attacks treated with study drug.

Exclusion Criteria:

* Any medical condition or clinical laboratory test which in the judgment of the Investigator makes the subject unsuitable for the study.
* Pregnant or breast-feeding women.
* Women of child-bearing potential not using or not willing to use highly effective contraception.
* Participant is at imminent risk of suicide (positive response to question 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS).
* Initiation of or a change in concomitant medication to reduce the frequency of migraine episodes since completing COL MIG-301/LAHJ (NCT02439320) or COL MIG-302/LAHK (NCT02605174).
* Participation in any clinical trial of an experimental drug or device since completing EoS/Visit 2 of COL MIG 301/LAHJ (NCT02439320) or COL MIG-302/LAHK (NCT02605174).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2171 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (194):
- United States (180):
  - Southview Medical Group, Birmingham, Alabama
  - Simon Williamson Clinic, Birmingham, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - East Valley Family Physicians, PLC, Chandler, Arizona
  - Radiant Research, Chandler, Arizona
  - Warner Family Practice, Chandler, Arizona
  - Fountain Hills Family Practice, P.C., Fountain Hills, Arizona
  - Neurological Physicians of Arizona Inc, Gilbert, Arizona
  - Thunderbird Internal Medicine, Glendale, Arizona
  - Thomas C. Lenzmeier, M.D., P.C, Glendale, Arizona
  - Central Arizona Medical Associates, PC, Mesa, Arizona
  - Desert Clinical Research, Mesa, Arizona
  - 21st Century Neurology, Phoenix, Arizona
  - Family Practice Specialists Ltd, Phoenix, Arizona
  - Central Phoenix Med Clinic LLC, Phoenix, Arizona
  - Thunderbird Internal Medicine, Phoenix, Arizona
  - Tatum Highlands Medical Associates, PLLC, Phoenix, Arizona
  - Radiant Research, Scottsdale, Arizona
  - Arizona Community Physicians, Tucson, Arizona
  - Orange Grove Family Practice, Tucson, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Radiant Research, Carlsbad, California
  - The Research Center of Southern California, Carlsbad, California
  - eStudySite, Chula Vista, California
  - Allied Clinical Research, Gold River, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Pacific Research Partners, LLC, Oakland, California
  - Desert Valley Research, Rancho Mirage, California
  - Northern California Clinical Research Center, Redding, California
  - Anderson Clinical Research, Redlands, California
  - California Research Foundation, San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Neurological Research Institute, Santa Monica, California
  - Radiant Research, Santa Rosa, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Encompass Clinical Research, Spring Valley, California
  - Radiant Research - Vista CA, Vista, California
  - Diablo Clinical Research, Walnut Creek, California
  - Mile High Primary Care, Aurora, Colorado
  - Alpine Clinical Research Center, Boulder, Colorado
  - Colorado Springs Family Practice, Colorado Springs, Colorado
  - Colorado Springs Health Partners, PC, Colorado Springs, Colorado
  - Clinical Trials of the Rockies, Denver, Colorado
  - Chase Medical Research, LLC, Hamden, Connecticut
  - Comprehensive Psychiatric Care, PC, Norwich, Connecticut
  - Nova Clinical Research, LLC, Bradenton, Florida
  - PAB Clinical Research, Brandon, Florida
  - Meridien Research, Brooksville, Florida
  - Avail Clinical Research LLC, DeLand, Florida
  - Clinical Research West Coast, Fort Myers, Florida
  - MD Clinical, Hallandale, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - Meridien Research, Maitland, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Prestige Clinical Research, Miami, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Florida Medical Center and Research, Inc., Miami, Florida
  - The Core Research Associates, Miami, Florida
  - Veritas Research Corp, Miami Lakes, Florida
  - Ocean Blue Medical Research Center, Inc., Miami Springs, Florida
  - Harmony Medical Research Institute, Inc, North Miami Beach, Florida
  - Clinical Neuroscience Solutions Inc, Orlando, Florida
  - Compass Research, Orlando, Florida
  - Radiant Research, Pinellas Park, Florida
  - Clinical Research Center, LLC, Royal Palm Beach, Florida
  - Meridien Research, St. Petersburg, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - Meridien Research, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Radiant Research, Atlanta, Georgia
  - Atlanta Center of Medical Research, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Urban Family Practice Associates, PC, Marietta, Georgia
  - Harbin Clinic, Rome, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Pinnacle Trials, Inc, Stockbridge, Georgia
  - Georgia Neurology & Sleep Medicine Associates, Suwanee, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Advanced Clinical Research LLC, Meridian, Idaho
  - Radiant Research, Chicago, Illinois
  - Michigan Avenue Internists, Chicago, Illinois
  - Medical and Procedural Specialists of Illinois, Chicago, Illinois
  - Evanston Premier Healthcare Research, LLC., Evanston, Illinois
  - Clinical Investigation Specialists Inc, Gurnee, Illinois
  - Synexus/Clinical Research Advantage, Evansville, Indiana
  - Synexus - US, Evansville, Indiana
  - Goldpoint Clinical Research LLC, Indianapolis, Indiana
  - Radiant Research, Inc., Council Bluffs, Iowa
  - Heartland Research Associates, Augusta, Kansas
  - Heartland Research Associates, Newton, Kansas
  - Continuum Health Care, Overland Park, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Central Kentucky Research Associates Inc, Lexington, Kentucky
  - Associates in Neurology, PSC, Lexington, Kentucky
  - Research Integrity, LLC, Owensboro, Kentucky
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Beacon Clinical Research, LLC, Quincy, Massachusetts
  - Michigan Head, Pain and Neurological Institute, Ann Arbor, Michigan
  - Radiant Research, Edina, Minnesota
  - Clinical Research Institute, Plymouth, Minnesota
  - West Florissant Internists, Bridgeton, Missouri
  - The Center For Pharmaceutical Research, Kansas City, Missouri
  - Radiant Research, St Louis, Missouri
  - Skyline Medical Center, Elkhorn, Nebraska
  - Prairie Fields Family Medicine, PC, Fremont, Nebraska
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Diagnostic Center of Medicine, Henderson, Nevada
  - Rita B. Chuang, MD LLC, Henderson, Nevada
  - Nevada Family Care, Henderson, Nevada
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Diagnostic Center of Medicine, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Regional Clinical Research, Endwell, New York
  - CNS Research Science, Inc., Jamaica, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Asheville Neurology Specialists, PA, Asheville, North Carolina
  - PMG Research of Cary, LLC, Cary, North Carolina
  - Radiant Research, Akron, Ohio
  - Synexus - US, Cincinnati, Ohio
  - IVA Research, Cincinnati, Ohio
  - Rapid Medical Research Inc, Cleveland, Ohio
  - Synexus - US, Columbus, Ohio
  - Oklahoma City Clinic, Edmond, Oklahoma
  - Oklahoma City Clinic, Midwest City, Oklahoma
  - Lynn Institute of Norman, Norman, Oklahoma
  - Oklahoma City Clinic, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Summit Research Network Inc, Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Partners in Clinical Research, LLC, Cumberland, Rhode Island
  - Lincoln Research, Lincoln, Rhode Island
  - West Bay Clinical Research, Warwick, Rhode Island
  - Primary Care Associates, Anderson, South Carolina
  - Radiant Research, Anderson, South Carolina
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Medical Research South, Charleston, South Carolina
  - Radiant Research, Greer, South Carolina
  - Mountain View Clinical Research, Inc., Greer, South Carolina
  - Coastal Carolina Research Center, Inc., Mt. Pleasant, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - Holston Medical Group Clinical Research, Kingsport, Tennessee
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Clinical Neuroscience Solutions Inc, Memphis, Tennessee
  - Nashville Neuroscience Group, Inc., Nashville, Tennessee
  - Central Texas Clinical Research, LLC, Austin, Texas
  - FutureSearch Trials, Austin, Texas
  - ACRC Trials, Austin, Texas
  - Tekton Research, Inc, Austin, Texas
  - ACRC Trials, Carrollton, Texas
  - FutureSearch Trials, Dallas, Texas
  - Radiant Research - Dallas North, Dallas, Texas
  - Protenium Clinical Research, Hurst, Texas
  - ACRC Trials, Plano, Texas
  - Doctors of Internal Medicine, Plano, Texas
  - Plano Internal Medicine Associates, Plano, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Radiant Research - San Antonio, San Antonio, Texas
  - MacGregor Medical Center, San Antonio, Texas
  - Ericksen Research and Development, Clinton, Utah
  - Radiant Research, Murray, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - J. Lewis Research, Inc., Salt Lake City, Utah
  - Jordan River Family Medicine, South Jordan, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Multicare Health System, Tacoma, Washington
  - Clinical Investigation Specialists Inc, Kenosha, Wisconsin
- Germany (4):
  - Synexus Clinical Research GmbH, Frankfurt am Main, Hesse
  - Gemeinschaftspraxis für Neurologie und Psychiatrie, Westerstede, Lower Saxony
  - Synexus Clinical Research GmbH, Leipzig, Saxony
  - Synexus Clinical Research GmbH, Berlin
- United Kingdom (10):
  - Synexus Ltd, Reading, Berkshire
  - Synexus Midlands Clinical Research Center, Edgbaston, Birmingham
  - Alverton Practice, Penzance, Cornwall
  - Kings College Hospital, London, Greater London
  - Synexus Manchester Clinical Research Centre, Manchester, Greater Manchester
  - Synexus Lancashire Clinical Research Centre, Chorley, Lancashire
  - Synexus Merseyside Clinical Research Centre, Waterloo, Merseyside
  - Synexus Hexham General Hospital, Hexham, Northumberland
  - Synexus Wales Clinical Research Centre, Cardiff, South Glamorgan
  - Synexus Scotland Clinical Research Centre, Glasgow, Strathclyde

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Blumenfeld A, Tepper SJ, Khanna R, Doty E, Vincent M, Miller SI. Serotonin syndrome in the acute treatment landscape of migraine: the lasmiditan experience. Front Neurol. 2023 Oct 27;14:1291102. doi: 10.3389/fneur.2023.1291102. eCollection 2023. PMID 37965170
- [Derived] Martin VT, Ahmed Z, Hochstetler HM, Baygani SK, Dong Y, Hauck PM, Khanna R. Tolerability and Safety of Lasmiditan Treatment in Elderly Patients With Migraine: Post Hoc Analyses From Randomized Studies. Clin Ther. 2021 Jun;43(6):1066-1078. doi: 10.1016/j.clinthera.2021.04.004. Epub 2021 Aug 6. PMID 34366152
- [Derived] Peres MFP, Vasudeva R, Baygani SK, Dennehy EB, Vincent M, Friedman DI. Lasmiditan efficacy in migraine attacks with mild vs. moderate or severe pain. Curr Med Res Opin. 2021 Jun;37(6):1031-1038. doi: 10.1080/03007995.2021.1903846. Epub 2021 Apr 7. PMID 33784930
- [Derived] Clemow DB, Hochstetler HM, Dong Y, Hauck P, Peres MFP, Ailani J. Effect of a change in lasmiditan dose on efficacy and safety in patients with migraine. Postgrad Med. 2021 May;133(4):449-459. doi: 10.1080/00325481.2020.1860619. Epub 2021 Mar 17. PMID 33730977
- [Derived] Smith T, Krege JH, Rathmann SS, Dowsett SA, Hake A, Nery ESM, Matthews BR, Doty EG. Improvement in Function after Lasmiditan Treatment: Post Hoc Analysis of Data from Phase 3 Studies. Neurol Ther. 2020 Dec;9(2):459-471. doi: 10.1007/s40120-020-00185-5. Epub 2020 May 23. PMID 32447545
- [Derived] Lipton RB, Lombard L, Ruff DD, Krege JH, Loo LS, Buchanan A, Melby TE, Buse DC. Trajectory of migraine-related disability following long-term treatment with lasmiditan: results of the GLADIATOR study. J Headache Pain. 2020 Feb 24;21(1):20. doi: 10.1186/s10194-020-01088-4. PMID 32093628
- [Derived] Brandes JL, Klise S, Krege JH, Case M, Khanna R, Vasudeva R, Raskin J, Pearlman EM, Kudrow D. Interim results of a prospective, randomized, open-label, Phase 3 study of the long-term safety and efficacy of lasmiditan for acute treatment of migraine (the GLADIATOR study). Cephalalgia. 2019 Oct;39(11):1343-1357. doi: 10.1177/0333102419864132. Epub 2019 Aug 21. PMID 31433669

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lasmiditan 100mg | Lasmiditan 200mg
Started | 1046 | 1125
Received at Least One Dose of Study Drug | 991 | 1039
Completed | 466 | 504
Not Completed | 580 | 621
Not completed — Adverse Event | 113 | 148
Not completed — Lost to Follow-up | 102 | 93
Not completed — Non-Compliance | 57 | 55
Not completed — Withdrawal by Subject | 229 | 214
Not completed — Physician Decision | 18 | 16
Not completed — Sponsor Request | 5 | 9
Not completed — Missing | 1 | 0
Not completed — Did Not Receive Study Drug | 55 | 86

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Lasmiditan 100mg: Participants received oral dose of 100mg Lasmiditan with in four hours of onset of migraine attack. If the migraine did not respond within 2 hours after first dose or if responded and recurred then a second dose was permitted within 24 hours after first dose.
- Total: Total of all reporting groups
Arm/Group | Lasmiditan 100mg | Lasmiditan 200mg | Total
Number analyzed (Participants) | 1046 | 1125 | 2171
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (12.25) | 43.4 (12.33) | 43.0 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All randomized participants with available gender data.
  Participants
    number analyzed (Participants) | 1046 | 1123 | 2169
    Female | 882 | 957 | 1839
    Male | 164 | 166 | 330
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 208 | 240 | 448
  Not Hispanic or Latino | 833 | 880 | 1713
  Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 11 | 15
  Asian | 7 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 4 | 6 | 10
  Black or African American | 203 | 194 | 397
  White | 805 | 884 | 1689
  More than one race | 11 | 14 | 25
  Unknown or Not Reported | 12 | 10 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1041 | 1065 | 2106
  United Kingdom | 5 | 38 | 43
  Germany | 0 | 22 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least 1 Treatment Emergent Adverse Event
Description: An AE with an onset on or within 48 hours after a dose of study drug, or an event that worsened in intensity within 48 hours of a dose of study drug was considered a treatment-emergent adverse event (TEAE).
  A summary of serious adverse events (SAEs) and other non-serious adverse events (AEs), regardless of causality, were reported in the Reported Adverse Events module.
Time Frame: Up to 12 months
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Lasmiditan 100mg | Lasmiditan 200mg
Number analyzed (Participants) | 991 | 1039
Participants | 447 | 545

2. Secondary Outcome: Percentage of Migraine Attacks With Pain Freedom (PF) at 2 Hours After Dose
Description: Pain freedom is defined as a reduction in headache severity from mild (1), moderate (2), or severe (3) at baseline to none (0).
Time Frame: Up to 12 months
Population: All randomized participants who treated at least 1 qualifying migraine attack within 4 hours of onset.
Measure: Number; unit: Percentage of PF Migraine Attacks
Units Other Than Participants: Migraine Attacks
Arm/Group | Lasmiditan 100mg | Lasmiditan 200mg
Number analyzed (Participants) | 954 | 1000
Number analyzed (Migraine Attacks) | 8837 | 8479
Percentage of PF Migraine Attacks | 26.7 | 32.2

3. Secondary Outcome: Percentage of Migraine Attacks With Most Bothersome Symptom-Free (MBS) at 2 Hours After Dose
Description: MBS-free, defined as the absence of the associated symptom of migraine (nausea, phonophobia, and/or photophobia) at 2 hours postdose that was identified predose as the most bothersome symptom.
Time Frame: Up to 12 months
Population: All randomized participants who treated at least 1 qualifying migraine attack within 4 hours of onset.
Measure: Number; unit: Percentage of MBS-Free Migraine Attacks
Units Other Than Participants: Migraine Attacks
Arm/Group | Lasmiditan 100mg | Lasmiditan 200mg
Number analyzed (Participants) | 954 | 1000
Number analyzed (Migraine Attacks) | 8045 | 7529
Percentage of MBS-Free Migraine Attacks | 37.2 | 40.8

4. Other Pre Specified Outcome: Percentage of Participants With Medical Resource Utilization
Description: Medical Resource utilization for any cardiovascular (CV) events and/or related resource utilization, such as visits to cardiologists, procedures, hospitalizations, new treatments or treatment adjustments for CV disease and any visits to an emergency room (ER) or physician's office for treatment of migraine was reported.
Time Frame: Up to 12 months
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Lasmiditan 100mg | Lasmiditan 200mg
Number analyzed (Participants) | 991 | 1039
Percentage of Participants
  Visit to cardiologist | 0.6 | 0.6
  Visit to primary care | 0.8 | 0.9
  Visit to Other providers | 0.1 | 0.2
  Hospitalized | 0.5 | 0.2
  Procedures performed | 0.8 | 0.6
  ER visits or visits to Physicians Office | 2.6 | 2.6

ADVERSE EVENTS:
Time Frame: Up to 12 Months
Description: All randomized participants who received at least one dose of study drug.
  Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | Lasmiditan 100mg | Lasmiditan 200mg
All-Cause Mortality (participants affected / at risk) | 0/991 | 0/1039
Serious Adverse Events (participants affected / at risk) | 29/991 | 36/1039
Other Adverse Events (participants affected / at risk) | 446/991 | 543/1039
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Lasmiditan 100mg (N=991) | Lasmiditan 200mg (N=1039)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (2) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Coccidioidomycosis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Relapsing-remitting multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3/845 (3) | 1/887 (1)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0/845 (0) | 1/887 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Schizoaffective disorder bipolar type (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0/845 (0) | 1/887 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0/845 (0) | 1/887 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0/845 (0) | 1/887 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Lasmiditan 100mg (N=991) | Lasmiditan 200mg (N=1039)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 3 (6) | 5 (5)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (3)
Diplacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (5)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 4 (4) | 4 (5)
Vertigo (Ear and labyrinth disorders) | 10 (15) | 24 (53)
Altered visual depth perception (Eye disorders) | 0 (0) | 1 (1)
Blindness transient (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Dyschromatopsia (Eye disorders) | 0 (0) | 2 (2)
Eye disorder (Eye disorders) | 0 (0) | 1 (3)
Iritis (Eye disorders) | 0 (0) | 1 (1)
Metamorphopsia (Eye disorders) | 0 (0) | 3 (3)
Miosis (Eye disorders) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 2 (2)
Photopsia (Eye disorders) | 3 (3) | 5 (6)
Strabismus (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 6 (8)
Visual impairment (Eye disorders) | 3 (7) | 8 (23)
Vitreous floaters (Eye disorders) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 6 (12)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 2 (3)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 39 (47) | 55 (81)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 4 (4) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 17 (18) | 11 (12)
Asthenia (General disorders) | 15 (38) | 24 (48)
Chest discomfort (General disorders) | 3 (64) | 4 (8)
Chills (General disorders) | 0 (0) | 3 (3)
Discomfort (General disorders) | 1 (1) | 3 (3)
Facial pain (General disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 47 (90) | 64 (159)
Feeling abnormal (General disorders) | 7 (11) | 8 (9)
Feeling cold (General disorders) | 1 (1) | 1 (3)
Feeling drunk (General disorders) | 2 (3) | 2 (4)
Feeling hot (General disorders) | 0 (0) | 3 (3)
Feeling jittery (General disorders) | 7 (9) | 5 (11)
Feeling of relaxation (General disorders) | 1 (2) | 1 (9)
Gait disturbance (General disorders) | 2 (3) | 4 (6)
Hunger (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 3 (5) | 2 (3)
Non-cardiac chest pain (General disorders) | 2 (2) | 4 (4)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Swelling face (General disorders) | 1 (1) | 2 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Sphincter of oddi dysfunction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (2)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0/845 (0) | 1/887 (1)
Body tinea (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 3 (3)
Influenza (Infections and infestations) | 2 (2) | 4 (4)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 9 (9)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4) | 8 (8)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 6 (6)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 5 (5)
Viral infection (Infections and infestations) | 2 (2) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (4) | 2 (2)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 1/845 (1) | 0/887 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 2 (3)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 2 (2) | 2 (2)
Blood triglycerides increased (Investigations) | 0 (0) | 2 (2)
Electrocardiogram t wave biphasic (Investigations) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 0 (0) | 2 (2)
Heart rate increased (Investigations) | 2 (2) | 1 (1)
Heart rate irregular (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Norovirus test positive (Investigations) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ligament laxity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (12) | 9 (17)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (7) | 6 (8)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 5 (6) | 7 (12)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 (23) | 16 (49)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/845 (1) | 0/887 (0)
Akathisia (Nervous system disorders) | 2 (3) | 2 (24)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 3 (11) | 7 (31)
Aura (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 7 (21) | 19 (31)
Cognitive disorder (Nervous system disorders) | 4 (5) | 3 (4)
Coordination abnormal (Nervous system disorders) | 0 (0) | 3 (4)
Disturbance in attention (Nervous system disorders) | 2 (2) | 6 (9)
Dizziness (Nervous system disorders) | 156 (336) | 220 (647)
Dysarthria (Nervous system disorders) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1) | 1 (1)
Fine motor skill dysfunction (Nervous system disorders) | 0 (0) | 3 (5)
Head discomfort (Nervous system disorders) | 1 (1) | 5 (7)
Headache (Nervous system disorders) | 3 (3) | 5 (5)
Hypersomnia (Nervous system disorders) | 2 (2) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 13 (16) | 21 (31)
Lethargy (Nervous system disorders) | 20 (36) | 14 (34)
Medication overuse headache (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 2 (3)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 9 (10) | 9 (9)
Mononeuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 53 (84) | 86 (293)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 5 (8) | 4 (5)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Sedation (Nervous system disorders) | 3 (9) | 5 (7)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (2)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Sleep paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 77 (153) | 95 (290)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Stupor (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Tarsal tunnel syndrome (Nervous system disorders) | 1 (2) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 8 (8) | 14 (19)
Visual field defect (Nervous system disorders) | 2 (2) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 4 (8) | 6 (23)
Affect lability (Psychiatric disorders) | 1 (2) | 0 (0)
Agitation (Psychiatric disorders) | 2 (3) | 1 (2)
Anxiety (Psychiatric disorders) | 8 (12) | 9 (9)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 3 (3)
Depersonalisation/derealisation disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 3 (3)
Disorientation (Psychiatric disorders) | 0 (0) | 8 (11)
Dysphoria (Psychiatric disorders) | 1 (1) | 3 (3)
Emotional distress (Psychiatric disorders) | 1 (1) | 0 (0)
Enuresis (Psychiatric disorders) | 1 (1) | 1 (1)
Euphoric mood (Psychiatric disorders) | 5 (7) | 11 (22)
Fear (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 5 (5) | 3 (3)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Hypnagogic hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 7 (10)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1)
Listless (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental fatigue (Psychiatric disorders) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (2) | 3 (7)
Panic attack (Psychiatric disorders) | 0 (0) | 3 (3)
Phonophobia (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 6 (7) | 5 (6)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/845 (0) | 1/887 (1)
Menstruation irregular (Reproductive system and breast disorders) | 1/845 (1) | 0/887 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal odour (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (5) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 3 (4)
Hot flush (Vascular disorders) | 3 (3) | 4 (5)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT02565186/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT02565186/SAP_001.pdf